CLINICAL TRIAL: NCT02017678
Title: A Single-arm, Open-label, Phase 2 Study of JX-594 (Thymidine Kinase-Deactivated Vaccinia Virus Plus GM-CSF) Administered by 5 Weekly Intravenous (IV) Infusions in Patients With Peritoneal Carcinomatosis of Ovarian Cancer Origin
Brief Title: Phase 2 Study of JX-594 in Patients With Peritoneal Carcinomatosis of Ovarian Cancer Origin
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Andrea McCart (Other)
Collaborators: Ontario Institute for Cancer Research (Other)
Responsible Party: Sponsor-Investigator, Andrea McCart, Gastrointestinal Surgical Oncologist, Mount Sinai Hospital, Canada
Organization: Mount Sinai Hospital, Canada (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZM-044
Record Dates: First submitted 2013-09-20; First posted 2013-12-23 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Ovarian Cancer
Keywords: JX-594; Ovarian cancer; Peritoneal; Carcinomatosis; Vaccinia virus; Oncolytic virus
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma; Vaccinia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- JX-594 IV Infusion (Experimental): Patients with peritoneal carcinomatosis of ovarian origin that are not eligible for curative treatments will receive 5 weekly IV infusions of JX-594
  Interventions: Biological: JX-594

INTERVENTIONS:
Biological: JX-594 — 5 weekly IV infusions of JX-594 followed by laparoscopy and biopsy on day 10 or 38.
  Other Names: vaccinia virus

SUMMARY:
This is a single-arm open-label Phase 2 study in patients with peritoneal carcinomatosis of ovarian origin that are not eligible for curative treatments. Patients will receive 5 weekly IV infusions of JX-594 until radiographically determined progressive disease. Patients will be allotted in a 1:1 ratio to undergo a laparoscopy and tumor biopsy 10 days after dose 1 or 10 days after Dose 5. Patients will be monitored on study until evidence of progression or death or for 12 months post treatment.

DETAILED DESCRIPTION:
This is a single-arm open-label Phase 2 study in patients with peritoneal carcinomatosis of ovarian origin that are not eligible for curative treatments. Patients will receive 5 weekly IV infusions of JX-594 and will continue to receive IV infusion of JX-594 every 3 weeks until radiographically determined progressive disease. Using a 2 stage trial design, if 2 or more of the first 15 patients show a clinical response as defined by Response Evaluation Criteria in Solid Tumors 1.10 criteria (or if 3 of the 15 have stable disease as defined by Modified Response Evaluation Criteria in Solid Tumors 1.1 or clinically), the arm will be expanded to a total of 25 patients (Stage 2).

In Stage 1, patients will be allotted in a 1:1 ratio to undergo a laparoscopy and tumor biopsy 10 days after dose 1 or 10 days after Dose 5. A decision as to whether laparoscopy will be performed in Stage 2 will be reached at the conclusion of Stage 1.

Patients will be monitored on study until evidence of progression or death or for 12 months post treatment

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed ovarian carcinomatosis with; no curative treatment options available, or the patient has refused or cannot tolerate the standard therapy. Patients must have had prior primary platinum based chemotherapy.
2. Radiologically evaluable disease.
3. At least 2 tumor masses amenable to biopsy (excisional or core) or laparoscopy. Tumor masses selected cannot be followed by Response Evaluation Criteria in Solid Tumors 1.1.
4. Expected survival ≥12 weeks
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
6. Women aged ≥18 years
7. Sexually active patients must be able and willing to abstain for a minimum of 15 days after treatment with JX-594 and subsequently use barrier method for at least 6 weeks after the last JX-594 treatment
8. Signed informed consent form
9. No contraindications to undergo general anesthetic or laparoscopy.
10. Laboratory requirements:

Hematology

* Absolute neutrophil count (ANC) ≥1.0 x 109/L
* Lymphocytes ≥0.5 x109/L
* Hemoglobin ≥90 g/L (correction with transfusion or erythropoietin based therapy allowed)
* Platelet count ≥75 x 109/L

Biochemistry

* Total bilirubin ≤1.5 x upper limit of normal (ULN)
* Alkaline Phosphatase (ALP), Aspartate transaminase (AST), alanine aminotransferase (ALT) ≤3 x ULN (if patient exhibits liver metastasis, up to 5 x ULN acceptable)
* Serum creatinine ≤1.5 x ULN or creatinine clearance is ≥1.0 mL/s according to Cockroft-Gault formula
* International normalized ratio (INR) ≤1.5 Serum chemistries within normal limits (WNL) or Grade 1 (with exception of sodium, potassium, glucose, calcium, phosphate,magnesium, chloride upon Investigator discretion)

Exclusion Criteria:

1. Significant immunodeficiency due to underlying illness (e.g., known HIV/AIDS) and/or medication (e.g., systemic corticosteroids taken for more than 4 weeks within the preceding 3 months). Intermittent doses of corticosteroids as an antiemetic for chemotherapy are acceptable. Patients have to be off continuous steroids for at least 4 weeks
2. Therapeutic anticoagulant therapy
3. History of severe exfoliative skin condition (e.g., eczema or ectopic dermatitis requiring systemic therapy for more than 4 weeks)
4. Tumor(s) invading a major vascular structure (e.g., carotid artery)
5. Clinically significant and uncontrolled pericardial or pleural effusions
6. Severe or unstable cardiac disease, including significant coronary artery disease (e.g., requiring angioplasty or stenting) within the preceding 12 months, unless well-controlled and on stable medical therapy for at least 3 months
7. Tumor burden >50% of abdominal cavity or malignant obstruction of small bowel or other condition that would preclude safe biopsy or laparoscopy
8. Brain metastasis: Viable central nervous system (CNS) malignancy associated with clinical symptoms (Note: enrollment allowed if completely resected or stable post radiotherapy >12 weeks).
9. Received anti-cancer therapy within 4 weeks prior to first treatment (6 weeks in case of mitomycin C or nitrosoureas)
10. Prior participation in other research protocol involving an investigational product within 4 weeks or 5 half-lives, whichever is longer, prior to first treatment
11. Medical condition, laboratory abnormality or active infection that in the judgment of the Principal Investigator may increase the risk associated with study participation or may prevent laparoscopy or may interfere with interpretation of study results and/or otherwise make the patient inappropriate for study entry
12. Use of interferon/pegylated interferon (PEG-IFN) or ribavirin that cannot be discontinued within 14 days prior to any JX-594 dose. (Note: please consult Ozmosis Research Inc. if patient is taking any other anti-viral medications to determine eligibility)
13. Unable to receive IV contrast for CT scanning due to documented history of iodinated contrast allergy unless controlled by medical intervention (e.g., premedication with steroids, diphenhydramine, or other anti-allergic medications)
14. Pregnant or nursing an infant
15. Pulse oximetry O2 saturation <90% at rest on room air
16. Experienced a severe systemic reaction or side-effect as a result of a previous smallpox vaccination.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Radiographic response of ovarian peritoneal carcinomatosis to JX-594 treatment | 6 weeks
  Determine radiographic response rate (response evaluation criteria in solid tumors [modified Response Evaluation Criteria in Solid Tumors 1.1])to JX-595

SECONDARY OUTCOMES:
Assessment of Adverse Events related to JX-594 administered by repetitive IV infusion | Weekly
  Collection of incidence(s) of treatment-emergent adverse events will be tabulated and stratified by severity and relationship to JX-594 administration
Response rate using modified immune criteria | 6 weeks
  Determine response rate using modified immune criteria in ovarian peritoneal carcinomatosis
Delivery of JX-594 in solid tumours | Weekly
  Determine the delivery of JX-594 to solid tumors after repetitive IV infusion in patients with peritoneal carcinomatosis
JX-594 Secondary Replication in blood over time | Weekly
  Determine the pharmacokinetics of JX-594 by examining secondary replication of viral genomes in blood over time.
Immune response to JX-594 | 6 weeks
  Determine the immune response to JX-594 by change in peripheral white blood cell counts over time
Response of tumour markers to JX-594 | Weekly
  Determine serum tumor marker response rate
Time to progressive disease | 6 weeks
  Determine time to progression of disease after JX-594 administration

CONTACTS AND LOCATIONS:
Overall Officials: Judith Andrea McCart, MD, Principal Investigator — MOUNT SINAI HOSPITAL; Helen MacKay, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Center, Toronto, Ontario, Canada